CLINICAL TRIAL: NCT05545124
Title: Clinical Study of Donafenib Combined With Tislelizumab in the Adjuvant Therapy of High-risk Recurrence-risk Primary Hepatocellular Carcinoma After Radical Surgical Resection
Brief Title: Study of Donafenib Combined With Tislelizumab in the Adjuvant Treatment of Primary HCC With High Risk of Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-388
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib+Tislelizumab (Experimental): Donafenib+Tislelizumab
  Interventions: Drug: Donafenib + Tislelizumab

INTERVENTIONS:
Drug: Donafenib + Tislelizumab — Donafenib 100mg, BID+Tislelizumab 200mg, D1; q3w

SUMMARY:
To explore the safety and preliminary efficacy of donafenib combined with tislelizumab in adjuvant therapy after radical surgical resection of primary hepatocellular carcinoma with high risk of recurrence.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, open-label clinical study. For HCC patients who the investigator believes can benefit from adjuvant treatment with donafenib combined with PD-1 monoclonal antibody, they will sign an informed consent form, and then start donafenib within 1-2 months after radical surgery (stable disease assessment or improvement). Adjuvant therapy with fenib combined with tislelizumab for 6 months, to explore the safety and efficacy of postoperative adjuvant therapy with donafenib combined with tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 years old (including the threshold value), male or female;
2. Received radical resection of liver cancer 4-8 weeks before enrollment;
3. Pathologically diagnosed as hepatocellular carcinoma and assessed by the investigator to have a high risk of recurrence;
4. No recurrence or metastasis was confirmed by imaging examination before enrollment;
5. Child-Pugh score of liver function A;
6. Eastern Cooperative Oncology Group (ECOG) physical status (PS) score of 0-1;
7. The expected survival period is not less than 3 months;
8. The doctor's decision to use Donafenib must be done before the patient is enrolled in the study;
9. For HBV-infected patients, if HBV-DNA is ≥104copies/ml within 14 days before enrollment, they should take antiviral treatment (entecavir is recommended), and then enter the study when it drops to <104copies/ml, and continue antiviral treatment and monitoring Liver function and serum HBV-DNA level;
10. Have sufficient organ functional reserve
11. Female patients with reproductive potential (referring to nonmenopausal or surgical sterilization), the serum pregnancy test results must be negative within 7 days before the administration of the study drug; female or male patients with reproductive potential, during the use of the study drug And within 60 days after the last dose, reliable contraceptive measures must be used;
12. Patients are voluntarily enrolled, can provide written informed consent, and can understand and comply with the experimental protocol, taking medication and follow-up.

Exclusion Criteria:

1. Pathologically diagnosed as mixed hepatocellular carcinoma-intrahepatic cholangiocarcinoma (HCC-ICC) or fibrolamellar hepatocellular carcinoma;
2. Past or current patients with congenital or acquired immunodeficiency diseases;
3. Active or previously recorded autoimmune diseases or inflammatory diseases, with vitiligo or asthma that has been completely resolved in childhood, without any intervention in adulthood can be included;
4. Combined with other liver diseases, including uncontrolled alcoholic hepatitis or other hepatitis, decompensated liver cirrhosis, severe fatty liver, hereditary liver disease, liver atrophy, superior vena cava syndrome, portal hypertension.
5. Have a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia found during chest CT scan screening;
6. Other malignancies within 5 years, unless the patient has received potentially curative treatment and there is no evidence of the disease within 5 years, but this time requirement (that is, within 5 years) does not apply to basal cell carcinoma of the skin that has been successfully resected , skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or other in situ carcinoma patients;
7. Have a history of serious mental illness in the past;
8. Suffering from diseases that affect the absorption, distribution, metabolism or clearance of the study drug (such as severe vomiting, chronic diarrhea, intestinal obstruction, malabsorption, etc.);
9. Received major surgery within 4 weeks before enrollment (determined by the investigator);
10. Patients who have received allogeneic stem cell or solid organ transplantation in the past, including patients after liver transplantation;
11. Received other anti-tumor systemic therapy before enrollment, including other traditional Chinese medicines with anti-tumor indications, less than 2 weeks or 5 drug half-lives (whichever is longer) after the completion of the treatment and before the drug in this study. , or patients whose adverse events caused by preoperative treatment did not recover to ≤CTCAE grade 1;
12. Received other adjuvant therapy after surgery (except antiviral therapy);
13. Systemic immunosuppressive drug therapy has been used within 2 weeks before enrollment, or systemic immunosuppressive drug therapy is expected to be required during the study period
14. Concomitant use of drugs that may prolong QTc and/or induce torsades de pointes (Tdp) or drugs that affect drug metabolism;
15. The patient is known or suspected to have a history of allergy to tyrosine kinase inhibitor (TKI) drugs and PD-1 drugs, or to the excipients of the study drug;
16. There is uncontrollable hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion;
17. Active bleeding or abnormal coagulation function, bleeding tendency or receiving thrombolysis, anticoagulation or antiplatelet therapy;
18. There is a history of gastrointestinal bleeding within the past 4 weeks or a clear tendency of gastrointestinal bleeding (such as: known local active ulcer lesions, fecal occult blood ++++ or above, such as persistent fecal occult blood+, gastroscopic examination should be performed), Or other conditions that may cause gastrointestinal bleeding as determined by the investigator (such as severe gastric fundus/esophageal varices);
19. Gastrointestinal perforation, abdominal fistula or abdominal abscess occurred within the past 6 months;
20. Thrombosis or thromboembolic events have occurred in the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.;
21. Cardiovascular disease with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within the past 6 months, congestive heart failure (NYHA classification > grade 2 of the New York Heart Association ), poorly controlled arrhythmias that require pacemaker therapy, and uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
22. Active infection;
23. Other significant clinical and laboratory abnormalities that the investigators consider to affect the safety evaluation, such as: uncontrolled diabetes mellitus, chronic kidney disease, peripheral neuropathy of grade II or above (CTCAE V5.0), abnormal thyroid function, etc.;
24. Have not recovered from surgery, such as unhealed incisions or serious postoperative complications;
25. Pregnant or breastfeeding women, as well as female or male patients with reproductive potential who are unwilling or unable to take effective contraceptive measures;
26. History of alcohol, psychotropic or other drug abuse within the past 6 months;
27. Received clinical trials of other drugs or medical devices within 4 weeks before enrollment;
28. Unable to follow the research protocol to receive treatment or follow up regularly;
29. Any other researchers who think that they cannot be included in the group

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival | 1 years
  Ratio of patients from first treatment to disease recurrence within 1 year

SECONDARY OUTCOMES:
recurrence-free survival with surgical resection | 2 years
  Time elapsed from surgical resection to tumor recurrence or death from any cause (if the subject died before disease recurrence)
overall survival | up to 1 years
  Time from enrollment date to date of death from any cause
adverse events | up to 1 years
  Incidence of adverse events in combination immunization with donafenib

CONTACTS AND LOCATIONS:
Overall Officials: Jinxue Zhou, Principal Investigator — Henan Cancer Hospital